CLINICAL TRIAL: NCT01319812
Title: The Treatment of Iliac and Femoral Atherosclerotic Lesions Using the Self-expanding Astron and Pulsar Stents
Brief Title: Investigational Device Exemption Study to Determine the Safety and Efficacy of the Astron and Pulsar Stents
Acronym: BIOFLEX-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOFLEX-I
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease
Keywords: Vascular intervention; Endovascular; Peripheral stent
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astron Stent Group (Experimental): Participants indicated for stenting in iliac atherosclerotic lesions.
  Intervention: Device: Astron Stents
  Interventions: Device: Astron Stents
- Pulsar Stent Group (Experimental): Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions.
  Intervention: Device: Pulsar Stents
  Interventions: Device: Pulsar Stents

INTERVENTIONS:
Device: Astron Stents — Implantation of self-expanding, bare-metal, nitinol stents for treatment of peripheral artery disease affecting the iliac artery.
  Other Names: Astron Stent
  Arms: Astron Stent Group
Device: Pulsar Stents — Implantation of self-expanding, bare-metal, nitinol stents for treatment of peripheral artery disease affecting superficial femoral or proximal popliteal arteries.
  Other Names: Astron Pulsar Stent; Pulsar-18 Stent; Pulsar Stent
  Arms: Pulsar Stent Group

SUMMARY:
The objective of this study is to separately demonstrate the safety and efficacy of BIOTRONIK's Astron and Pulsar stents. The Pulsar stent will be used for the treatment of femoro-popliteal lesions, located in the native superficial femoral artery (SFA) or proximal popliteal artery (PPA), while the Astron stent will be used for the treatment of the common or external iliac artery lesions.

ELIGIBILITY:
Inclusion Criteria

To support the objectives of this study, the following initial inclusion criteria must be met for a subject to be enrolled and considered for the index procedure:

* Age ≥ 18 years
* Willingness to comply with study follow-up requirements
* Candidate for PTA
* Life-style limiting claudication or rest pain with an ABI ≤ 0.9 (resting or exercise). Thigh brachial index (TBI) may be used / performed if ABI is inadequate.
* Written informed consent

For a subject to receive an investigational stent, the following procedure-related criteria must be met:

* One de novo, restenotic or occluded lesion representing a femoro-popliteal or iliac indication OR Two de novo, restenotic or occluded lesions representing one femoro-popliteal indication and one iliac indication on contralateral limbs - (i.e. one lesion per limb)
* Lesions may be one solid lesion or a series of multiple, smaller lesions to be treated as one lesion
* Subjects with bilateral, SFA/PPA disease (i.e. one SFA/PPA lesion per limb) are eligible for enrollment into the study. The target lesion will be selected at the investigator's discretion based on study eligibility criteria. The contralateral SFA/PPA intervention may be performed at the time of the index procedure (prior to treatment of study lesion); however, the use of an investigational treatment is prohibited. If the contralateral SFA/PPA intervention is not performed at the time of the index procedure, the intervention must be performed at least 30 days after the index procedure. The use of an investigational treatment for the contralateral intervention is prohibited.
* Subjects with bilateral, iliac disease (i.e. one iliac lesion per limb) are eligible for enrollment into the study. The target lesion will be selected at the investigator's discretion based on study eligibility criteria. The contralateral iliac intervention may be performed at the time of the index procedure; however, the use of an investigational treatment is prohibited. If the contralateral iliac intervention is not performed at the time of the index procedure, the intervention must be performed at least 30 days after the index procedure. The use of an investigational treatment for the subsequent contralateral intervention is also prohibited.
* Femoro-popliteal lesions must be located at least 1 cm distal to the profunda femoris artery and at least 3 cm above the knee joint (radiographic joint space)
* Iliac lesions must be located only in either the common or external iliac artery
* Lesions must be treatable with a maximum of two stents
* Angiographic evidence of ≥ 70% stenosis or occlusion (operator visual assessment)
* Lesion length ≤ 190 mm (if de novo or restenotic) or ≤ 100 mm (if occluded)
* Target vessel reference diameter: 2.5 to 6 mm (SFA/PPA) or 6 to 9 mm (iliac arteries) by visual estimate
* Angiographic evidence of patent SFA and PPA (iliac indication) and angiographic evidence of at least one distal vessel runoff to the foot (both femoro-popliteal and iliac indications). Patent is defined as < 50% stenosis.
* For SFA/PPA intervention, a significant stenosis (> 70%) or occlusion of an ipsilateral, inflow artery (e.g. aortoiliac, common femoral) must be successfully treated (use of investigational treatment prohibited) just prior to treatment of the target lesion. Successful treatment is defined as no complications and less than 30% residual stenosis following intervention.

Exclusion Criteria

To support the objectives of this study, the following initial exclusion criteria must not be present for a subject to be enrolled:

* Subjects pregnant or planning to become pregnant during the course of the study
* Life expectancy of less than one year
* Rutherford-Becker category 5 or 6. Subjects with ulcers caused by venous disease may be enrolled in the study.
* Previously stented lesion(s) in the target vessel
* Target lesion(s) received previous treatment within 30 days prior to enrollment
* Prior peripheral vascular bypass surgery involving the target limb(s)
* Thrombophlebitis or deep vein thrombosis within the past 30 days
* Known allergy to nitinol (nickel and/or titanium)
* Participation in any other clinical investigational device or drug study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.
* Previous stroke or transient ischemic attack within the last three months prior to enrollment
* Previous coronary or peripheral bypass surgery (non-target limb) within 30 days prior to enrollment
* Intolerance to contrast agents that cannot be medically managed and/or intolerance to anti-platelet, anti-coagulant or thrombolytic medications
* Refuses blood transfusions
* Any medical condition, that in the opinion of the investigator, poses an unacceptable risk for implant of a stent according to the study indications

For a subject to receive an investigational stent the following procedure-related criteria must not be present:

* INR ≥ 1.6
* Concomitant renal failure with serum creatinine level > 2.5 mg/dL
* Unresolved neutropenia (white blood cell count < 3,000 / µL) or thrombocytopenia (platelet count < 80,000 / µL) at the time of the index procedure
* Unresolved bleeding disorder (INR ≥ 1.6) at the time of the index procedure
* Presence of other ipsilateral, arterial lesions distal to the target lesion requiring treatment within 30 days of the index procedure (either before or after) or at the time of the index procedure
* Additional percutaneous interventional procedures (cardiac and/or peripheral) planned within 30 days after the index procedure
* Presence of a complication following pre-dilation of target lesion
* Presence of a target vessel/lesion that is excessively tortuous or calcified or is adjacent to an acute thrombus that is unresponsive to anti-thrombotic therapies
* Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion
* Target lesion requires the use of cutting balloons, atherectomy or ablative devices
* Subjects with less than single vessel runoff to the foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burket, MD, Principal Investigator — University of Toledo
Locations (34):
- United States (32):
  - Fremont, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Rockford, Illinois
  - Munster, Indiana
  - Houma, Louisiana
  - Lansing, Michigan
  - Saginaw, Michigan
  - Wyoming, Michigan
  - Ypsilanti, Michigan
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Ridgewood, New Jersey
  - New York, New York
  - The Bronx, New York
  - Gastonia, North Carolina
  - High Point, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Camp Hill, Pennsylvania
  - Doylestown, Pennsylvania
  - Langhorne, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Rock Hill, South Carolina
  - Kingsport, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - McKinney, Texas
  - Tyler, Texas
  - Waco, Texas
- Canada (2):
  - Montreal
  - Toronto

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Burket MW, Brodmann M, Metzger C, Tan K, Jaff MR. Twelve-Month Results of the Nitinol Astron Stent in Iliac Artery Lesions. J Vasc Interv Radiol. 2016 Nov;27(11):1650-1656.e1. doi: 10.1016/j.jvir.2016.06.008. Epub 2016 Aug 16. PMID 27542591

RESULTS

PARTICIPANT FLOW:
Groups:
- Astron Stent Group: Subjects implanted with an Astron stent.
- Pulsar Stent Group: Subjects implanted with an Astron Pulsar or Pulsar-18 stent.
Period: Overall Study
Arm/Group | Astron Stent Group | Pulsar Stent Group
Started | 161 | 302
Completed | 145 | 280
Not Completed | 16 | 22

BASELINE CHARACTERISTICS:
Population: The two arms of the BIOFLEX-I study were distinct with no overlap. Totals present here were automatically generated by the clinicaltrials.gov system. Four participants were enrolled in both the Astron and Pulsar stent groups, as allowed in the study protocol. Therefore any presented totals may not be accurate aggregates of data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Astron Stent Group | Pulsar Stent Group | Total
Number analyzed (Participants) | 161 | 302 | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (10.1) | 67.3 (10.3) | NA (NA) — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 97 | 153
  Male | 105 | 205 | 310
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 143 | 281 | 424
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 22 | 26
  White | 152 | 273 | 425
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 91 | 187 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Canada | 38 | 29 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Austria | 32 | 34 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Belgium | 0 | 32 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Switzerland | 0 | 6 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Germany | 0 | 14 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Medical History [Number; unit: Participants]
  Diabetes | 32 | 123 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Hypertension | 117 | 255 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Hyperlipidemia | 125 | 245 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Current smoker | 78 | 122 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Smoked within last 5 years | 36 | 46 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Never smoked or not within last 5 years | 47 | 134 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Cerebrovascular disease | 22 | 48 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  History of congestive heart failure | 11 | 27 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  History of ischemic heart disease | 69 | 124 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  History of coronary revasularization | 54 | 110 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Renal insufficiency | 11 | 17 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Lesion Location [Number; unit: Participants]
  Common iliac | 107 | 0 | 107
  External iliac | 54 | 0 | 54
  Ostial SFA | 0 | 2 | 2
  Proximal SFA | 0 | 38 | 38
  Mid SFA | 0 | 156 | 156
  Distal SFA | 0 | 99 | 99
  Proximal popliteal | 0 | 7 | 7
Lesion Calcification [Number; unit: Participants]
  None | 47 | 82 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Moderate | 68 | 91 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Severe | 46 | 129 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Lesion Length [Mean (Standard Deviation); unit: mm] | 35.9 (21.3) | 82.0 (46.9) | NA (NA) — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Vessel Diameter [Mean (Standard Deviation); unit: mm]
  Pre-deployment Minimum Lumen Diameter (MLD) | 2.1 (1.3) | 1.0 (0.9) | NA (NA) — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Post-deployment Minimum Lumen Diameter (MLD) | 6.0 (1.2) | 4.1 (0.7) | NA (NA) — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  Reference vessel diameter | 7.6 (1.5) | 5.0 (0.9) | NA (NA) — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Distal Vessel Runoff [Number; unit: Participants]
  Not Available | 35 | 32 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  0 Vessel | 9 | 19 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  1 Vessel | 32 | 74 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  2 Vessel | 48 | 93 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
  3 Vessel | 37 | 84 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
Trans-Atlantic Inter-Society Consensus (TASC II) Type [Number; unit: Participants] — TASC II grading is from the Trans-Atlantic Inter-Society Consensus. Type A lesions include a single stenosis <10 cm long or a single occlusion <5cm long; type B lesions include multiple lesions <5 cm, a single lesion <15cm, or a single popliteal stenosis; type C lesions include multiple stenosis or occlusions >15 cm with or without calcification, or a chronic total occlusion >20cm involving the popliteal; type D lesions include chronic total occlusions of the popliteal artery and proximal vessels. Generally, Type D lesions are mores severe than Type A lesions.
  Participants
    Type A | 99 | 166 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
    Type B | 56 | 106 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
    Type C | 6 | 26 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.
    Type D | 0 | 3 | NA — Study arms are independent with no overlap or comparison. A total would not present meaningful information and would be conflated by four subjects who were enrolled in both arms of the study.

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Endpoint for the Pulsar Stent: Primary Patency
Description: The primary effectiveness endpoint for the Pulsar stent group is the primary patency rate at 12 months post-index procedure. Primary patency is defined as freedom from more than 50% restenosis based on the duplex ultrasound peak systolic velocity ratio, comparing data within the treated segment to the proximal normal segment or based on a clinically-indicated TLR with angiographic evidence of > 50% stenosis.
Time Frame: 12 months
Population: Participants for whom patency could be confirmed at 12 months.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pulsar Stent Group: Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions.
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 268
Percentage of participants | 66.8 [60.8 to 72.4]

2. Primary Outcome: Safety Endpoint for the Pulsar Stent: Freedom From Procedure- or Stent-related Major Adverse Events
Description: The primary safety endpoint for the Pulsar stent is the freedom from procedure- or stent-related major adverse events at 30 days post-index procedure. The major adverse event rate includes mortality, target lesion revascularization and index limb amputation.
Time Frame: 30 days
Population: All participants implanted with an Astron Pulsar or Pulsar-18 stent.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 302
Percentage of participants | 99.7 [98.2 to 100.0]

3. Primary Outcome: Safety and Effectiveness Endpoint for the Astron Stent - Percentage of Participants With Major Adverse Events (MAE)
Description: The primary endpoint for the Astron stent is a composite of the rate of procedure- or stent-related major adverse events at 12 months post-index procedure. The major adverse event rate includes 30-day mortality, along with 12-month rates of target lesion revascularization and index limb amputation. Success was measured against a performance goal of 15%, given a 7.5% expected 12-month MAE rate, with an assumed delta value of 7.5%.
Time Frame: 12 months
Population: Includes all participants who underwent successful implantation and either met the 30-day mortality categorization or completed a 12-month evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Astron Stent Group: Participants indicated for stenting in iliac atherosclerotic lesions.
Arm/Group | Astron Stent Group
Number analyzed (Participants) | 146
Percentage of participants | 2.1 [0.4 to 5.9]

4. Primary Outcome: Percentage of Participants With Primary Safety Endpoint (Post Market Analysis)
Description: Freedom from a composite of clinically-driven target lesion revascularization (TLR) and index limb amputation at 36 months.
Time Frame: 36 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 257
percentage of participants | 78.2 [72.7 to 83.1]

5. Secondary Outcome: Secondary Safety Assessment for the Pulsar Stent: Individual Rates of Mortality, TLR, and Index Limb Amputation
Description: Evaluate the contribution of the individual rates of mortality, target lesion revascularization (TLR) and index limb amputation at 30 days post-index procedure to the primary safety endpoint for the Pulsar stent.
Time Frame: 30 days
Population: All participants implanted with an Astron Pulsar or Pulsar-18 stent.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 302
Percentage of participants
  Freedom from 30 day mortality | 99.7 [98.2 to 100.0]
  Freedom from 30 day TLR | 100.0 [98.8 to 100.0]
  Freedom from 30 day index limb amputation | 100.0 [98.8 to 100.0]

6. Secondary Outcome: Long-Term Safety Assessment for the Pulsar Stent: Major Adverse Event Rate
Description: Evaluate the long-term major adverse event rate of the Pulsar stent. Likewise, the endpoint will evaluate the contribution of the individual rates of 30-day mortality and 12-month target lesion revascularization and index limb amputation rates to this overall, long-term major adverse event rate.
Time Frame: 12 months
Population: Participants who reached at least 395 calendar days post procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 283
Percentage of participants
  30-day mortality | 0.4 [0.0 to 2.0]
  Target lesion revascularization | 12.4 [8.8 to 16.8]
  Index limb amputation | 0.4 [0.0 to 2.0]

7. Secondary Outcome: Stent Integrity Assessment for the Pulsar Stent: Stent Fracture Rate
Description: Evaluate the Pulsar stent integrity as measured by x-ray at 12 months post-index procedure. An independent angiographic core laboratory reviewed x-ray imaging for presence or absence of a stent fracture. Fractures were assessed with Grade I indicating a single tine fracture, Grade II indicating multiple tine fracture, Grade III indicating stent fracture(s) with preserved alignment of the components, Grade IV indicating stent fracture(s) with mal-alignment of the components, and Grade V stent fracture(s) in a trans-axial spiral configuration. Generally, fractures of Grade I are least severe, increasing in severity to Grade V.
Time Frame: 12 months
Population: Participants with 12 month (395 day) diagnostic X-ray available for fracture evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 243
Participants
  Overall stent fracture at 12 months | 14
  Grade I stent fracture at 12 months | 4
  Grade II stent fracture at 12 months | 3
  Grade III stent fracture at 12 months | 3
  Grade IV stent fracture at 12 months | 4
  Grade V stent fracture at 12 months | 0

8. Secondary Outcome: Secondary Safety Assessment for the Astron Stent - Distribution of MAE Rate
Description: Evaluate the contribution of the individual rates of 30-day mortality and 12-month target lesion revascularization and index limb amputation rates to the primary endpoint for the Astron stent.
Time Frame: 12 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group
Number analyzed (Participants) | 146
Percentage of participants
  30-day mortality | 0.7 [0.0 to 3.8]
  Target Lesion Revascularization | 1.4 [0.2 to 4.5]
  Index limb amputation | 0.0 [0.0 to 2.5]

9. Secondary Outcome: Secondary Effectiveness Assessment for the Astron Stent - Primary Patency Rate
Description: Evaluate the primary patency of the Astron stent at 12 months post-index procedure as measured by duplex ultrasound. Primary patency is defined as freedom from more than 50% restenosis based on the duplex ultrasound peak systolic velocity ratio, comparing data within the treated segment to the proximal normal segment or based on a clinically-indicated TLR with angiographic evidence of > 50% stenosis.
Time Frame: 12 months
Population: Includes all participants who underwent successful implantation and had a 12-month evaluable duplex ultrasound assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group
Number analyzed (Participants) | 128
Percentage of participants | 89.8 [83.3 to 94.5]

10. Secondary Outcome: Secondary Effectiveness Assessment for the Astron and Pulsar Stents - Primary Assisted Patency
Description: Evaluate the primary assisted patency rate (freedom from remote Target Vessel Revascularization [TVR]) for the Astron and Pulsar stent at 12 months post-index procedure.
Time Frame: 12 months
Population: Includes all participants who underwent successful implantation and were included in the 12-month ITT analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 146 | 275
Percentage of participants | 97.9 [94.1 to 99.6] | 98.9 [96.8 to 99.8]

11. Secondary Outcome: Secondary Effectiveness Assessment for the Astron and Pulsar Stents - Secondary Patency
Description: Evaluate the secondary patency rate (freedom from bypass and amputation of the target limb) for the Astron and Pulsar stent at 12 months post-index procedure.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 146 | 276
Percentage of participants | 99.3 [96.2 to 100.0] | 98.2 [95.8 to 99.4]

12. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Ankle - Brachial Index (ABI) Measurement
Description: The purpose of this endpoint is to compare the ABI measurements between baseline and 12 months post-index procedure. ABI is the ratio of systolic blood pressure of ankle relative to systolic blood pressure of arm.
Time Frame: 12 months
Population: Analysis conducted on paired data. ABI measurements were available for 141 participants from both baseline and the 12-month visit for the Astron stent group. ABI measurements were available for 266 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Ratio (ABI score)
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 141 | 266
Ratio (ABI score)
  Baseline ABI | 0.71 (0.15) | 0.70 (0.14)
  12-Month Visit ABI | 0.94 (0.18) | 0.91 (0.19)
  ABI difference | 0.23 (0.19) | 0.22 (0.21)

13. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Six-Minute Walk Test
Description: The purpose of this endpoint is to compare the distance walked during the 6-minute walk test between baseline and 12 months post-index procedure.
Time Frame: 12 months
Population: Analysis conducted on paired data. Six-minute walk test results were available for 131 participants from both baseline and the 12-month visit for the Astron stent group. Six-minute walk test results were available for 247 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 131 | 247
Feet
  Six-minute walk distance at baseline | 868.9 (446.5) | 875.3 (379.1)
  Six-minute walk distance at 12-month visit | 1026.4 (469.5) | 1088.9 (468.9)
  Six-minute walk distance difference | 157.5 (420.6) | 213.6 (412.7)

14. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Walking Impairment Questionnaire PAD Specific Score
Description: The purpose of this endpoint is to compare Walking Impairment Questionnaire (WIQ) Peripheral Arterial Disease (PAD) specific score between baseline and 12 months post-index procedure. The WIQ is a subjective questionnaire completed by participants at baseline and the 12 month visit which asks questions about mobility to assess walking impairment. Larger numbers indicate better outcomes, with a minimum score of 0 and a maximum score of 100. Please see the following publication for further information:
  Hiatt WR, Hirsch AT, Regensteiner JG, et al. Clinical Trials for Claudication. Assessment of Exercise Performance, Functional Status, and Clinical Endpoints. Vascular Clinical Trialists. Circulation. 1995;92:614-621
Time Frame: 12 months
Population: Analysis conducted on paired data. WIQ PAD responses were available for 143 participants from both baseline and the 12-month visit for the Astron stent group. WIQ PAD responses were available for 265 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Units on a scale (WIQ score)
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 143 | 265
Units on a scale (WIQ score)
  WIQ PAD Specific Score at Baseline | 36.2 (29.0) | 36.7 (28.1)
  WIQ PAD Specific Score at 12-Month Visit | 80.1 (29.2) | 75.8 (32.3)
  WIQ PAD Specific Score Difference | 43.9 (36.8) | 39.1 (40.4)

15. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Walking Impairment Questionnaire Walking Distance Score
Description: The purpose of this endpoint is to compare Walking Impairment Questionnaire Walking Distance score between baseline and 12 months post-index procedure. The WIQ is a subjective questionnaire completed by participants at baseline and the 12 month visit which asks questions about mobility to assess walking impairment. Larger numbers indicate better outcomes, with a minimum score of 0 and a maximum score of 100.. Please see the following publication for further information:
  Hiatt WR, Hirsch AT, Regensteiner JG, et al. Clinical Trials for Claudication. Assessment of Exercise Performance, Functional Status, and Clinical Endpoints. Vascular Clinical Trialists. Circulation. 1995;92:614-621
Time Frame: 12 months
Population: Analysis conducted on paired data. WIQ walking distance scores were available for 144 participants from both baseline and the 12-month visit for the Astron stent group. WIQ walking distance scores were available for 264 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Units on a scale (WIQ score)
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 144 | 264
Units on a scale (WIQ score)
  WIQ Walking Dist Score at Baseline | 21.3 (24.2) | 26.1 (26.3)
  WIQ Walking Dist Score at 12-Month Visit | 62.0 (39.5) | 58.7 (38.9)
  WIQ Walking Dist Score Difference | 40.7 (38.0) | 32.6 (37.4)

16. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Walking Impairment Questionnaire Walking Speed Score
Description: The purpose of this endpoint is to compare Walking Impairment Questionnaire Walking Speed score between baseline and 12 months post-index procedure. The WIQ is a subjective questionnaire completed by participants at baseline and the 12 month visit which asks questions about mobility to assess walking impairment. Larger numbers indicate better outcomes, with a minimum score of 0 and a maximum score of 100.. Please see the following publication for further information:
  Hiatt WR, Hirsch AT, Regensteiner JG, et al. Clinical Trials for Claudication. Assessment of Exercise Performance, Functional Status, and Clinical Endpoints. Vascular Clinical Trialists. Circulation. 1995;92:614-621
Time Frame: 12 months
Population: Analysis conducted on paired data. WIQ walking speed scores were available for 143 participants from both baseline and the 12-month visit for the Astron stent group. WIQ walking speed scores were available for 263 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Units on a scale (WIQ score)
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 143 | 263
Units on a scale (WIQ score)
  WIQ Walking Speed Score at Baseline | 22.3 (19.2) | 25.2 (21.2)
  WIQ Walking Speed Score at 12-Month Visit | 43.8 (28.6) | 43.5 (28.0)
  WIQ Walking Speed Score Difference | 21.5 (27.5) | 18.3 (28.1)

17. Secondary Outcome: Functional Assessments for Subjects With the Astron and Pulsar Stents - Walking Impairment Questionnaire Stair Climbing Score
Description: The purpose of this endpoint is to compare Walking Impairment Questionnaire Stair Climbing score between baseline and 12 months post-index procedure. The WIQ is a subjective questionnaire completed by participants at baseline and the 12 month visit which asks questions about mobility to assess walking impairment. Larger numbers indicate better outcomes, with a minimum score of 0 and a maximum score of 100. Please see the following publication for further information:
  Hiatt WR, Hirsch AT, Regensteiner JG, et al. Clinical Trials for Claudication. Assessment of Exercise Performance, Functional Status, and Clinical Endpoints. Vascular Clinical Trialists. Circulation. 1995;92:614-621
Time Frame: 12 months
Population: Analysis conducted on paired data. WIQ stair climbing scores were available for 142 participants from both baseline and the 12-month visit for the Astron stent group. WIQ stair climbing scores were available for 255 participants from both baseline and the 12-month visit for the Pulsar stent group.
Measure: Mean (Standard Deviation); unit: Units on a scale (WIQ score)
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 142 | 255
Units on a scale (WIQ score)
  WIQ Stair Climbing Score at Baseline | 30.0 (27.1) | 36.8 (31.5)
  WIQ Stair Climbing Score at 12-Month Visit | 56.1 (36.8) | 56.9 (37.8)
  WIQ Stair Climbing Score Difference | 26.1 (35.6) | 20.1 (36.0)

18. Secondary Outcome: Acute Procedural Success for Astron and Pulsar Stent
Description: Evaluate the acute procedural success of the Astron and Pulsar stent. Acute procedural success is defined as completion of the assigned procedure, the stented lesion having less than 30% residual stenosis determined by angiography immediately after stent placement and no MAEs before hospital discharge.
Time Frame: 30 days
Population: Includes all participants who underwent implantation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 161 | 302
Percentage of participants | 95.0 [90.4 to 97.8] | 98.0 [95.7 to 99.3]

19. Secondary Outcome: Clinical Success
Description: Evaluate the 30-day clinical success of the procedure. The 30-day clinical success is defined as completion of the assigned procedure, the stented lesion having less than 30% residual stenosis determined by angiography immediately after stent placement and no MAEs within 30 days of the index procedure.
Time Frame: 30 days
Population: The Astron stent group includes all participants who underwent implantation. The Pulsar stent group includes all participants who underwent implantation except for one, due to subject death occurring in the first 30 days.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 161 | 301
Percentage of participants | 95.0 [90.4 to 97.8] | 97.7 [95.3 to 99.1]

20. Secondary Outcome: Secondary Safety Assessment for Astron and Pulsar Stent: Adverse Event Rates
Description: Evaluate the rates of all individual adverse event types that are not included in the primary endpoint analyses for the Astron stent and the Pulsar stent group. Please see the Serious Adverse Events and Other Adverse Events sections for event details.
Time Frame: 12 month
Population: Includes all participants who underwent implantation.
Measure: Number; unit: Participants with event
Arm/Group | Astron Stent Group | Pulsar Stent Group
Number analyzed (Participants) | 161 | 302
Participants with event
  Serious adverse events | 67 | 180
  Non-serious adverse events | 94 | 277

21. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - 30 Day MAE Rate
Description: Compare the 30 day MAE rate results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: 30 days
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Groups:
- Astron Stent Group - Occlusive Lesion: Participants indicated for stenting in iliac atherosclerotic lesions where the target lesion was occlusive (100% stenosis).
- Astron Stent Group - Non-occlusive: Participants indicated for stenting in iliac atherosclerotic lesions where the target lesion was non-occlusive (70% to 99% stenosis).
- Pulsar Stent Group - Occlusive Lesion: Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions where the target lesion was occlusive (100% stenosis).
- Pulsar Stent Group - Non-occlusive Lesion: Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions where the target lesion was non-occlusive (70% to 99% stenosis).
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 12 | 134 | 91 | 211
Percentage of participants | 0.0 | 2.2 | 0.0 | 0.5

22. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - Primary Patency at 12-months
Description: Compare the primary patency at 12-months results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 10 | 118 | 82 | 186
Percentage of participants | 80.0 | 90.7 | 59.8 | 69.9

23. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - Primary Assisted Patency at 12-Months
Description: Compare the primary assisted patency (freedom from remote TVR) at 12-months results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 12 | 134 | 83 | 192
Percentage of participants | 100.0 | 97.8 | 96.4 | 100.0

24. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - Secondary Patency Rate at 12-Months
Description: Compare the secondary patency (freedom from bypass and amputation of the target limb) at 12-months results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 12 | 134 | 84 | 192
Percentage of participants | 100.0 | 99.3 | 97.6 | 98.4

25. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - Acute Procedure Success
Description: Compare the acute procedure success results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: Acute / Date of Procedure
Population: Includes all participants who underwent implantation.
Measure: Number; unit: Percentage of participants
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 13 | 148 | 91 | 211
Percentage of participants | 100.0 | 94.6 | 97.8 | 98.1

26. Secondary Outcome: Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar Stent - 30-Day Clinical Success
Description: Compare the 30-day clinical success results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar stent group.
Time Frame: 30 days
Population: Includes all participants who underwent implantation.
Measure: Number; unit: Percentage of participants
Arm/Group | Astron Stent Group - Occlusive Lesion | Astron Stent Group - Non-occlusive | Pulsar Stent Group - Occlusive Lesion | Pulsar Stent Group - Non-occlusive Lesion
Number analyzed (Participants) | 13 | 148 | 90 | 211
Percentage of participants | 100.0 | 94.6 | 97.8 | 97.6

27. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - MAE Rate
Description: Compare the MAE rate results between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Groups:
- Pulsar Stent Group - Standard Lesion Length: Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions with a lesion length between 20 mm and 140 mm.
- Pulsar Stent Group - Long Lesion Length: Participants indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions with a lesion length between 141 mm and 190 mm.
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 247 | 36
Percentage of participants | 10.9 | 25.0

28. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - Primary Patency at 12 Months
Description: Compare the primary patency rate at 12 months between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 235 | 33
Percentage of participants | 68.5 | 54.5

29. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - Stent Fracture Rate at 12 Months
Description: Compare the stent fracture rate at 12 months between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 213 | 30
Percentage of participants | 4.7 | 13.3

30. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - Primary Assisted Patency at 12 Months
Description: Compare the primary assisted patency rate at 12 months between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 241 | 34
Percentage of participants | 99.2 | 97.1

31. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - Secondary Patency Rate at 12 Months
Description: Compare the secondary patency rate at 12 months between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 12 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 239 | 34
Percentage of participants | 98.8 | 94.1

32. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - Acute Procedure Success
Description: Compare the acute procedure success results between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: Acute / Date of Procedure
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 265 | 37
Percentage of participants | 98.1 | 97.3

33. Secondary Outcome: Comparison of Endpoint Results Between Standard and Long Lesions for the Pulsar Stent - 30-day Clinical Success
Description: Compare the 30-day clinical success results between evaluable subjects treated with standard length lesions (between 20 mm and 140 mm) and evaluable subjects treated for long lesions (between 141 mm and 190 mm) for the Pulsar stent group.
Time Frame: 30 days
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsar Stent Group - Standard Lesion Length | Pulsar Stent Group - Long Lesion Length
Number analyzed (Participants) | 265 | 36
Percentage of participants | 97.7 | 97.2

34. Secondary Outcome: Number of Participants With Freedom From Clinically-driven TLR and Index Limb Amputation at 24 Months (Post Approval)
Description: Evaluate the rate of freedom from target lesion revascularization (TLR) and/or index limb amputation for the Pulsar stent.
Time Frame: 24 Months
Population: Evaluable participants for TLR at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 268
Participants | 217

35. Secondary Outcome: Safety Assessment for the Pulsar Stent: Percentage of Participants With Mortality, TLR, and Index Limb Amputation (Post Approval)
Description: as for outcome 5
Time Frame: 24 Months
Population: Evaluable participants at 24 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 269
percentage of participants
  MAE - Related to stent or index procedure | 19.3 [14.8 to 24.6]
  30-day mortality | 0.4 [0.0 to 2.1]
  Clinically-driven TLR | 19.0 [14.5 to 24.2]
  Index limb amputation | 0.8 [.01 to 2.7]

36. Secondary Outcome: Percentage of Participants for the Pulsar Stent Group With MAE (30-day Mortality, Clinically-driven TLR, and Index Limb Amputation) and Their Components at 36 Months (Post Approval).
Description: Evaluate the MAE rate and the individual component rates of mortality at 30 days post-index procedure, target lesion revascularization (TLR) and index limb amputation for the Pulsar stent.
Time Frame: 36 Months
Population: Evaluable participants at 36 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 258
percentage of participants
  MAE - Related to stent or index procedure | 22.1 [17.2 to 27.7]
  - 30-day mortality | 0.4 [0.0 to 2.1]
  - Clinically-driven TLR | 21.8 [16.9 to 27.3]
  - Index limb amputation | 1.2 [0.2 to 3.4]

37. Secondary Outcome: Percentage of Participants With Target Lesion Revascularization (TLR) at 24 Months (Post Approval) (Pulsar Stent Group)
Time Frame: 24 Months
Population: Evaluable participants for TLR at 24 months.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 268
percentage of Participants | 20.9 [16.2 to 26.3]

38. Secondary Outcome: Percentage of Participants With Target Lesion Revascularization (TLR) at 36 Months (Post Approval) (Pulsar Stent Group)
Time Frame: 36 Months
Population: Evaluable participants for TLR at 36 months. Pulsar Stent Group Post Market Analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 257
percentage of participants | 23.7 [18.7 to 29.4]

39. Secondary Outcome: Number of Participants With Stent Fracture at 24 Months (Post Approval).
Time Frame: 24 Months
Population: Evaluable participants for stent fracture at 24 months. Pulsar Stent Group Post Market Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 230
Participants | 10

40. Secondary Outcome: Number of Participants With Stent Fracture at 36 Months (Post Approval) (Pulsar Stent Group).
Time Frame: 36 Months
Population: Evaluable participants for stent fracture at 36 months. Pulsar Stent Group Post Market Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 204
Participants | 13

41. Secondary Outcome: Percentage of Subjects With Serious Adverse Events at 36 Months (Post Approval) (Pulsar Stent Group).
Description: Summary of serious adverse event rates at 36 months. Refer to SAE section.
Time Frame: 36 months
Population: Pulsar Stent Group Post Market Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsar Stent Group
Number analyzed (Participants) | 302
Participants | 230

ADVERSE EVENTS:
Time Frame: Enrollment through 12-months post-procedure for Astron group Serious and Non-serious Adverse Events. Enrollment through 36-months post-procedure for Pulsar group Serious and Non-serious Adverse Events.
Description: For non-serious adverse events with 0 listed for Astron, there may have been events reported for the category however the number events did not reach the 5% threshold for reporting.
Groups:
- Astron Stent Group: Subjects indicated for stenting in iliac atherosclerotic lesions.
- Pulsar Stent Group: Subjects indicated for stenting in superficial femoral or proximal popliteal atherosclerotic lesions.
Arm/Group | Astron Stent Group | Pulsar Stent Group
All-Cause Mortality (participants affected / at risk) | 5/161 | 27/302
Serious Adverse Events (participants affected / at risk) | 67/161 | 180/302
Other Adverse Events (participants affected / at risk) | 33/161 | 179/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astron Stent Group (N=161) | Pulsar Stent Group (N=302)
Abnormal coagulation profile (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 12 (15)
Bleeding requiring treatment (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal aortic aneurysm (Cardiac disorders) | 0 (0) | 2 (2)
Angina (Cardiac disorders) | 1 (1) | 8 (9)
Atrial arrhythmia (Cardiac disorders) | 2 (2) | 9 (10)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 9 (9)
Cardiac catheterization (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 11 (12)
Coronary artery disease (Cardiac disorders) | 4 (4) | 26 (27)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1) | 2 (2)
Dyspnea (Cardiac disorders) | 0 (0) | 6 (6)
Edema (Cardiac disorders) | 0 (0) | 4 (4)
Elevated troponin (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (Cardiac disorders) | 0 (0) | 1 (1)
Fluctuating blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
Heart block (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 7 (8)
Hypertensive crisis (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 9 (12)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Medication reaction/toxicity (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 14 (16)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Patent foramen ovale closure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Superior mesenteric artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 7 (8)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Valvular heart disease (Cardiac disorders) | 0 (0) | 5 (5)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Worsening cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Worsening coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Worsening heart failure (Cardiac disorders) | 1 (1) | 18 (24)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 6 (7)
Hyperlipidemia (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 6 (6)
Worsening diabetic control (Endocrine disorders) | 0 (0) | 4 (4)
Bleeding left eye (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 6 (6)
Horner's syndrome, right eye (Eye disorders) | 0 (0) | 1 (1)
Neovascular glaucoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 5 (6)
Bariatric surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding (Gastrointestinal disorders) | 5 (5) | 10 (17)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon/rectal polyp(s) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonoscopy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 5 (6)
Gallstone (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric bypass surgery (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer(s) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia, hiatal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia, inguinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ischemic colitis/colon polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea and/or vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6)
Suspected abdominal ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ventral and umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death-cause undetermined (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 4 (5)
Fever (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 4 (4)
Open or non-healing wound/ulcer (General disorders) | 0 (0) | 2 (2)
Open wounds due to injury (General disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 2 (2)
Traumatic injury (General disorders) | 1 (1) | 6 (6)
Weakness (General disorders) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Breast (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5)
Cellulitis (Infections and infestations) | 0 (0) | 6 (7)
Clostridium difficile (Infections and infestations) | 0 (0) | 2 (2)
E. coli infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Fungemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Groin wound (Infections and infestations) | 0 (0) | 1 (1)
Infection resulting in amputation (Infections and infestations) | 0 (0) | 1 (1)
Ingrown toenail (Infections and infestations) | 0 (0) | 1 (1)
Inner ear infection (Infections and infestations) | 0 (0) | 1 (1)
MRSA (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis resulting in amputation (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 17 (17)
Pocket infection (Infections and infestations) | 0 (0) | 1 (1)
Positive E. faecalis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 5 (6)
Septic shock resulting in amputation (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Surgical site - elbow (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Toenail fungus (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 8 (8)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound drainage/Purulant drainage (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Allergic reaction to contrast media or anti-thrombotic meds (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Anaphylactic shock (Injury, poisoning and procedural complications) | 0 | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chronic shoulder dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (11)
Gonathrosis of the knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar laminectomy and fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 14 (16)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 19 (21)
Vocal cord polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Axonal sensible polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 1 (1) | 8 (9)
Tinnitus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 2 (2) | 3 (3)
Vasovagal episode (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Altered mental status (Psychiatric disorders) | 1 (1) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystocele (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Increased serum creatinine (Renal and urinary disorders) | 0 (0) | 3 (3)
Kidney stone(s) (Renal and urinary disorders) | 0 (0) | 5 (5)
Muliple organ failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 6 (8)
Ureter obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Worsening renal function (Renal and urinary disorders) | 0 (0) | 9 (9)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hernia vaginal (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Profound hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory compromise (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sudden respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin condition/rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Angioplasty on left external iliac and SFA (Surgical and medical procedures) | 1 (1) | 0 (0)
Failure to deliver stent to intended site (Surgical and medical procedures) | 1 (1) | 1 (1)
Hematoma (Surgical and medical procedures) | 0 (0) | 5 (5)
ICD/pacemaker device replacement (Surgical and medical procedures) | 1 (1) | 2 (2)
Nausea and/or vomiting (Surgical and medical procedures) | 0 (0) | 1 (1)
Planned carotid stenting (Surgical and medical procedures) | 0 (0) | 1 (1)
Planned PVI in contralateral extremity (Surgical and medical procedures) | 0 (0) | 10 (10)
Post-surgical wound discomfort (Surgical and medical procedures) | 0 (0) | 1 (1)
Pseudoaneurysm - procedure related (Surgical and medical procedures) | 0 (0) | 3 (3)
Thrombosis or occlusion during stenting procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Vessel dissection or perforation during placement of thrombolysis catheter (Surgical and medical procedures) | 0 (0) | 1 (1)
Vessel dissection or perforation during PTA/ prior to stenting (Surgical and medical procedures) | 1 (1) | 8 (8)
Vessel dissection or perforation during stenting procedure (Surgical and medical procedures) | 1 (1) | 4 (4)
Acute mesenteric ischemia (Vascular disorders) | 0 (0) | 1 (1)
Arterial embolization distal to puncture site (Vascular disorders) | 0 (0) | 1 (1)
Basilar artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Carotid artery disease (Vascular disorders) | 0 (0) | 1 (1)
Carotid stenosis (Vascular disorders) | 0 (0) | 11 (13)
Compartment syndrome (Vascular disorders) | 0 (0) | 1 (1)
Contralateral iliac dissection (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Discoloration of 5th right toe (Vascular disorders) | 0 (0) | 1 (1)
Gangrene resulting in amputation (Vascular disorders) | 0 (0) | 2 (2)
Hematoma - non-index procedure related (Vascular disorders) | 0 (0) | 7 (7)
Numbness and/or tingling in lower extremities (Vascular disorders) | 0 (0) | 1 (1)
Occlusion of bypass graft left illiopopliteal bypass conduit (Vascular disorders) | 1 (1) | 0 (0)
Open or non-healing wound/ulcer (Vascular disorders) | 0 (0) | 7 (8)
Peripheral ischemia (Vascular disorders) | 3 (4) | 3 (3)
Phlegmon of the forefoot - led to amputation (Vascular disorders) | 0 (0) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 3 (3) | 3 (3)
Pseudoaneurysm - non-index procedure related (Vascular disorders) | 0 (0) | 2 (2)
Renal artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Right femoral occlusion (Vascular disorders) | 2 (2) | 0 (0)
Stenosis or occlusion in contralateral extremity (Vascular disorders) | 14 (15) | 66 (83)
Stenosis or occlusion in target extremity outside of stent segment (Vascular disorders) | 8 (9) | 50 (69)
Stenosis or occlusion of target lesion within stent segment (Vascular disorders) | 2 (2) | 61 (84)
Subclavian stenosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis in target lesion stenosis/ occlusion (Vascular disorders) | 0 (0) | 6 (7)
Thrombosis of a non-target vessel, contralateral (Vascular disorders) | 0 (0) | 1 (1)
Thrombotic occlusion of a bypass graft (Vascular disorders) | 0 (0) | 2 (2)
Varicose veins (Vascular disorders) | 0 (0) | 2 (2)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Worsening claudication (Vascular disorders) | 0 (0) | 2 (2)
Worsening of claudication (Vascular disorders) | 1 (1) | 2 (2)
Worsening of PAD (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astron Stent Group (N=161) | Pulsar Stent Group (N=302)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 16 (17)
Chest pain (Cardiac disorders) | 8 (11) | 24 (26)
Dizziness/ lightheadedness (Cardiac disorders) | 8 (8) | 17 (20)
Dyspnea (Cardiac disorders) | 0 (0) | 23 (26)
Edema (Cardiac disorders) | 0 (0) | 33 (38)
Hypertension (Cardiac disorders) | 0 (0) | 22 (25)
Leg pain and/or cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 16 (17)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 (24) | 67 (96)
Numbness and/or tingling in lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 16 (17)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 19 (23)
Skin condition/rash (Skin and subcutaneous tissue disorders) | 0 (0) | 16 (20)
Hematoma - Non-index procedure related (Surgical and medical procedures) | 0 (0) | 24 (27)
Stenosis or occlusion in contralateral extremity (Vascular disorders) | 0 (0) | 39 (46)
Stenosis or occlusion in target exremity outside of stent segment (Vascular disorders) | 0 (0) | 23 (27)
Stenosis or occlusion of target lesion within stent segment (Vascular disorders) | 0 (0) | 39 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No